CLINICAL TRIAL: NCT07065656
Title: Study of High-velocity Nasal Insufflation Versus Non-invasive Positive Pressure Ventilation for Emergency Type 2 Respiratory Failure: a Non-inferiority Randomized Controlled Trial (The SHINE Trial)
Brief Title: HVNI vs NIPPV in Type 2 Respiratory Failure
Acronym: SHINE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Vapotherm, Inc. (Industry)
Responsible Party: Principal Investigator, Mui Teng Chua, Asst Prof Mui Teng Chua, National University Hospital, Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHINE
Record Dates: First submitted 2025-06-21; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Failure; Hypoxia; Hypercapnia
MeSH Terms: conditions — Respiratory Insufficiency; Hypoxia; Hypercapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Experimental): In the HVNI group, patients will be given oxygen therapy via the Vapotherm high velocity therapy (HVT) 2.0 (Vapotherm, Inc, Exeter, NH) using a small-bore cannula, with a flow rate of up to 45 L/min, starting temperature of 37oC and FiO2 of up to 1.0. Adjustments in flow, temperature and FiO2 will be up to the attending physician's discretion to alleviate respiratory distress and optimize comfort.
  Interventions: Device: Vapotherm high velocity therapy (HVT) 2.0 (Vapotherm, Inc, Exeter, NH)
- Control (Active Comparator): For the NIPPV group, ventilation will be performed with the Respironics Vision V60 (Philips Healthcare, Murrysville, PA) using an oronasal mask of appropriate size, with FiO2 (up to 1.0), inspiratory (IPAP 12 to 20 cmH2O) and expiratory (EPAP 5 to 10 cm H2O) pressures titrated to alleviate patient's respiratory distress.
  Interventions: Device: Respironics Vision V60

INTERVENTIONS:
Device: Vapotherm high velocity therapy (HVT) 2.0 (Vapotherm, Inc, Exeter, NH) — Oxygen therapy will be given via the Vapotherm high velocity therapy (HVT) 2.0 (Vapotherm, Inc, Exeter, NH) using a small-bore cannula, with a flow rate of up to 45 L/min, starting temperature of 37oC and FiO2 of up to 1.0.
  Arms: Intervention
Device: Respironics Vision V60 — Ventilation will be performed with the Respironics Vision V60 (Philips Healthcare, Murrysville, PA) using an oronasal mask of appropriate size, with FiO2 (up to 1.0), inspiratory (IPAP 12 to 20 cmH2O) and expiratory (EPAP 5 to 10 cm H2O) pressures titrated to alleviate patient's respiratory distress.
  Arms: Control

SUMMARY:
The purpose of this study is to determine if high velocity nasal insufflation (HVNI) is comparable to non-invasive positive pressure ventilation (NIPPV) in treatment of emergency patients with acute respiratory acidosis. In our non-inferiority trial, we hypothesize that HVNI is inferior to NIPPV in reducing PaCO2 in type 2 respiratory failure (T2RF) due to any cause by a pre-specified non-inferiority margin of 4.3% decrease in PaCO2 levels after 30 minutes of treatment. The primary aim is to evaluate if HVNI is non-inferior to NIPPV in reducing PaCO2 levels in patients with T2RF from any cause. Eligible patients will be randomized to HVNI (intervention) or NIPPV (control).

DETAILED DESCRIPTION:
Acute respiratory and cardiac conditions are frequently encountered in the emergency department (ED), varying from mild to severe. Among the critically ill, up to one-third of them may have respiratory failure at presentation. Prompt and effective intervention in the ED can reduce adverse patient outcomes, decrease hospital length of stay and need for intubation, and limit resource utilization. Common conditions seen in the ED that can result in respiratory failure include acute pulmonary edema, acute exacerbation of chronic obstructive pulmonary disease (COPD), asthma, pneumonia, restrictive lung disease and bronchiectasis. Traditionally, NIPPV has been the modality of choice in management of hypercapnic respiratory failure in COPD and cardiogenic pulmonary edema. It provides positive pressure to the airways, helping to improve ventilation and reduce the work of breathing by assisting with both inspiration and expiration. It is, however, associated with side effects and complications such as pneumothorax, nasal bridge skin abrasions, claustrophobia, patient intolerance due to the positive pressure or dry and non-humidified air, gastric distension, aspiration and ill-fitting masks resulting in air leaks and eventual therapeutic failure. Additionally, patients are unable to speak or eat during application of the NIPPV mask and suctioning of oral secretions is also precluded. In the event of treatment failure with NIPPV, the next treatment modality would inadvertently be endotracheal intubation, which has its short-term risks such as peri-intubation hypotension and cardiac arrest, and longer-term risk of ventilator-associated pneumonia.

High flow nasal oxygenation (HFNO) is a relatively new modality for treating patients with respiratory failure and it involves delivering oxygen to patients using a specialized device to provide a high flow (up to 60 L/min) of warm, humidified oxygen far beyond the maximum of 4 to 6 L/min by standard nasal cannula. The benefits of HFNO include higher patient tolerance and comfort compared to NIPPV, no interruption in oxygen therapy during eating, reducing metabolic work in heating and air humidification, easy to use and monitor, and avoiding the complications associated with intubation and mechanical ventilation. Risks of skin abrasions and aspiration associated with NIPPV can also be prevented. A variety of devices exists. One variant is high velocity nasal insufflation (HVNI), which utilizes a smaller bore nasal cannula to flush airways and improve oxygenation. At the same flow rate, HVNI generates a higher nasopharyngeal pressure with a higher flow velocity than HFNO and is more effective in washing out extra-thoracic dead space,8 potentially more effective than HFNO in reducing PaCO2 levels.

The focus on HFNO has predominantly been on oxygenation rather than ventilation and the few studies on T2RF mostly focused on patients with COPD. Additionally, current evidence in HVNI use for acute hypercapnia is still lacking. Therefore, our study aims to evaluate if HVNI is non-inferior to NIPPV in reducing PaCO2 levels in acute T2RF from any cause. If proven to be non-inferior, this could be an alternative therapy for patients with respiratory acidosis, especially if they are unable to tolerate NIPPV or developed complications from it, thereby reducing the need for intubation and its potential adverse effects in such patients.

Specific aims & hypothesis

The purpose of this study is to determine if high velocity nasal insufflation (HVNI) is comparable to non-invasive positive pressure ventilation (NIPPV) in treatment of emergency patients with acute respiratory acidosis. In our non-inferiority trial, we hypothesize that HVNI is inferior to NIPPV in reducing PaCO2 in type 2 respiratory failure (T2RF) due to any cause by a pre-specified non-inferiority margin of 4.3% decrease in PaCO2 levels after 30 minutes of treatment. Our specific aims are as follows:

1. Primary aim: To evaluate if HVNI is non-inferior to NIPPV in reducing PaCO2 levels in patients with T2RF from any cause
2. Secondary aims: To compare if HVNI is similar to NIPPV in terms of treatment failure or need for intubation, and if HVNI can improve respiratory rate and patient's comfort level, and reduce adverse events associated with NIPPV

Randomization will be performed in random permutated variable blocks of 4 and 6. The block lengths will be kept unknown to the study team as per ICH E9 guideline. However, block randomization will ensure the numbers in each group will remain similar throughout the study, should we fail to recruit the targeted number of patients. Allocation concealment will be maintained until the registration and randomization process is completed.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged 21 years and above, who require NIPPV for T2RF due to any cause in the Emergency Medicine Department of the National University Hospital

Exclusion Criteria:

* patients with "do-not-resuscitate" orders that include NO non-invasive ventilation use [patients with max NIV status will still be included]
* clinical suspicion or confirmed diagnosis of base of skull fractures or severe facial trauma that precludes NIPPV or nasal cannula placement
* vulnerable patient populations (e.g., pregnant women, prisoners)
* patients who refused consent
* hemodynamic instability (e.g., hypotension requiring immediate resuscitation), cardiac or respiratory arrest
* patients who require emergency intubation

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in PaCO2 levels at 30 and 60 minutes | 30 minutes and 60 minutes
  Change in PaCO2 levels obtained on ABG results 30 minutes and 60 minutes after start of HVNI or NIPPV [baseline ABG and ABGs at 30 minutes and 60 minutes will be performed]

SECONDARY OUTCOMES:
Change in RR | 30 minutes and 60 minutes
  Change in respiratory rate 30 minutes and 60 minutes after initiation of HVNI or NIPPV
Change in dypsnea level | 30 minutes and 60 minutes
  Change in Modified Borg dyspnea scale 30 minutes and 60 minutes after initiation of HVNI or NIPPV
Proportion of treatment failure | Duration of therapy in emergency department, an average of 4 hours
  Proportion of treatment failure (defined as need to convert to another oxygenation/ventilation therapy by clinical or ABG results, and need for intubation)
Adverse events | Duration of therapy in emergency department, an average of 4 hours
  Adverse events due to therapy rendered e.g., facial pain due to NIPPV mask application, vomiting, aspiration